CLINICAL TRIAL: NCT00218322
Title: Atomoxetine in Adolescents With Attention Deficit Hyperactivity Disorder (ADHD) and Substance Use Disorder (SUD)
Brief Title: Effectiveness of ATMX in Treating Adolescents With ADHD and SUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Timothy Wilens, MD, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-16264-1; K24DA016264 (NIH); K24-16264-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Substance-Related Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Treatment with placebo or atomoxetine for 12 weeks.
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Atomoxetine hydrochloride

INTERVENTIONS:
Drug: Atomoxetine hydrochloride — Atomoxetine up to maximum dose of 40 to 100mg/day in daily dosing based on body weight up to 12 weeks of the study.
  Arms: 2
Drug: Placebo — Placebo up to maximum dose of 40 to 100mg/day in daily dosing based on body weight up to 12 weeks of the study.
  Arms: 1

SUMMARY:
Adolescents with attention deficit hyperactivity disorder (ADHD) often develop substance use disorders (SUD). The purpose of this study is to evaluate the effectiveness of atomoxetine in treating adolescents dually diagnosed with ADHD and SUD.

DETAILED DESCRIPTION:
High rates of ADHD have been reported in adolescents with SUD. In addition, untreated ADHD is a risk factor for developing SUD. Atomoxetine is a norepinephrine reuptake inhibitor, and is currently used to treat adolescents with ADHD. The purpose of this trial is to evaluate the efficacy of atomoxetine in treating adolescents dually diagnosed with ADHD and SUD.

This study will last up to 18 weeks. Participants will receive six treatments of manual-driven, cognitive behavioral therapy for substance abuse over at 6 or earlier weeks. Participants and their parents will partake in therapy sessions. Subjects who have completed at least 2 weeks of CBT will be eligible to enter the controlled trial, at which point participants will be randomly assigned to receive either atomoxetine or placebo, which they will take once daily for 12 weeks. At the Week 12 study visit, participants will be assessed for symptoms of ADHD and SUD.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of ADHD
* Current or recent (within the three months prior to study entry) SUD, including marijuana and alcohol abuse
* ADHD CGI-S score of greater to or equal to 4

Exclusion Criteria:

* Any Unstable medical condition
* Recent history of intravenous drug use or cocaine dependence
* Currently abusing ecstasy, cocaine, gamma-hydroxybutyrate, methamphetamine, amphetamine, opioids, phencyclidine, or benzodiazepine
* Mental retardation or organic brain syndrome
* Currently psychotic or history of bipolar disorder
* Currently taking any psychotropic or anti-substance abuse disorder medications
* Current DSM-IV diagnosis of major depression, depressive disorder, or anorexia
* Pregnant or breastfeeding

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2004-09; Primary Completion 2006-03 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Symptoms of ADHD and SUD (measured at Week 12) | 12 Weeks (LOCF)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E. Wilens, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States